CLINICAL TRIAL: NCT00354627
Title: Early Access of TMC125 in Combination With Other Antiretrovirals in Treatment-experienced HIV-1 Infected Subjects With Limited Treatment Options
Brief Title: The TMC125-C214 Study Provides Early Access to TMC125 for HIV-1 Infected Patients Who Have Failed Multiple Antiretroviral Regimens and Will Also Gather Information on the Long-term Safety and Tolerability of TMC125 Combined With Other Antiretroviral Drugs
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR002743; TMC125-C214 (Other: Tibotec Pharmaceuticals, Ireland); NCT00613236 (obsolete NCT alias)
Record Dates: First submitted 2006-07-18; First posted 2006-07-20 (Estimated); Last update posted 2015-06-12 (Estimated); Status verified 2015-06

CONDITIONS: HIV-1
Keywords: HIV-1; Early Access Program (EAP); TMC125; treatment-experienced; failing multiple antiretroviral (ARV) regimens; limited to no treatment options
MeSH Terms: interventions — etravirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TMC125 (Experimental): TMC125 200 mg b.i.d. till commercially available.
  Interventions: Drug: TMC125

INTERVENTIONS:
Drug: TMC125 — 200 mg b.i.d. till commercially available.

SUMMARY:
The purpose of this study is to provide early access of TMC125 to HIV-1 infected patients who have failed multiple antiretroviral (ARV) regimens. Information on safety and tolerability aspects of TMC125 in combination with other ARVs in treatment-experienced HIV-1 patients with limited treatment options will be assessed. Available data regarding the effectiveness of the drug will also be collected. To be eligible, patients should be failing their current ARV regimen or be on a treatment interruption, should have previously received 2 different protease inhibitor (PI) containing regimens and be at least 3-class experienced (protease inhibitors [PI], nucleoside/tide reverse transcriptase inhibitors [N[t]RTIs] and non-nucleoside reverse transcriptase inhibitors [NNRTIs]) or at least 2-class experienced (PIs and N[t]RTIs) with primary NNRTI resistance. TMC125 will be administered in combination with an investigator-selected background of additional ARVs from the list of allowed medications.

DETAILED DESCRIPTION:
This is an open label trial with primary objective to provide early access to TMC125 for treatment-experienced HIV-1 infected patients who have failed multiple antiretroviral (ARV) regimens and have limited treatment options with currently approved ARVs. The secondary objective of this trial is to gather information on the safety and tolerability aspects of TMC125 in combination with other ARVs. Available efficacy data will also be collected. Patients should be at least 3-class experienced or 2-class experienced with primary non-nucleoside reverse transcriptase inhibitor (NNRTI) resistance. They should also have previously received 2 different protease inhibitor-based regimens (low-dose ritonavir is not counted as a protease inhibitor (PI) regimen), be on a treatment interruption or not be virologically suppressed on their current regimen, and not be able to use currently approved NNRTIs due to resistance (primary or acquired) and/or intolerance. Patients must also meet all in- and exclusion criteria. TMC125 (200mg twice daily) will be provided once the patient has been confirmed eligible for entry. Once treatment with TMC125 in combination with other ARVs has been initiated, patients must be instructed to follow the recommended visit schedule based on routine clinical care. Safety and tolerability of the entire antiretroviral therapy (ART) regimen, including TMC125, should be monitored by the investigator as per standard clinical practice. However, it is recommended that visits be planned 4 and 12 weeks following initiation of TMC125 in combination with other ARVs and every 12 weeks thereafter while on therapy during this trial. Adverse events (AEs) leading to treatment interruption or discontinuation and all serious adverse events (SAEs), with the exception of Acquired Immunodeficiency Syndrome (AIDS) defining illnesses (CDC class C) unless fatal or considered to be related to TMC125, will be collected. Other adverse events will be collected only if required as per local regulations. The background ARVs may be changed at any time during the trial, at the discretion of the investigator due to the development of resistance, intolerance, toxicity, etc. while continuing treatment with TMC125 if in the investigator's assessment the patient still benefits from treatment with TMC125. If changes in the background regimen are made, it is recommended that a follow-up visit be planned 4 weeks after the change in therapy. Treatment with investigational medication will be continued until virologic failure, treatment-limiting toxicity, subject lost to follow-up, patient's withdrawal, pregnancy, discontinuation of TMC125 development or when TMC125 has become commercially available in the patient's country. Patients will be instructed to orally take two 100 mg tablets of TMC125 following a meal every 12 hours. TMC125 (200 mg twice daily) must be used in combination with other antiretroviral drugs. Treatment with investigational medication will continue until virologic failure, treatment-limiting toxicity, patient lost to follow-up, withdrawal, pregnancy, discontinuation of TMC125 development or when TMC125 becomes commercially available in the patient's country.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 3-class experienced (3 classes of licensed oral antiretrovirals: nucleoside/tide reverse transcriptase inhibitors [N[t]RTI], protease inhibitors [PI], non-nucleoside reverse transcriptase inhibitors [NNRTI])
* Patients with primary NNRTI resistance can be included if they are experienced with at least 2 classes of ARVs (PIs, N[t]RTIs) and meet all the other inclusion criteria
* Patient has previously received 2 different PI-based regimens
* Patient is unable to use currently approved NNRTIs due to resistance (primary or acquired) and/or intolerance
* Patient, if currently receiving an ARV regimen, is not achieving adequate virologic suppression on his/her current regimen.

Exclusion Criteria:

* Prior or current participation in DUET trials (TMC125-C206 or TMC125-C216).
* Use of disallowed concomitant therapy, including disallowed antiretrovirals (ARV)
* Use of investigational ARVs (with exceptions)
* Any active clinically significant disease (e.g., cardiac dysfunction, pancreatitis, acute viral infection) or findings during screening of medical history or physical examination that is not either resolved or stabilized for at least 30 days before the Screening Phase
* Pregnant or breast-feeding female
* Female patient of childbearing potential not using effective non-hormonal birth control methods
* Patients with specific laboratory abnormalities
* Patients with clinical or laboratory evidence of significantly decreased hepatic function or decompensation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5178 (Actual)
Dates: Start 2006-01; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
The primary objective of TMC125-C214 is to provide early access to TMC125 for treatment-experienced HIV-1 infected patients who have failed multiple antiretroviral (ARV) regimens and have limited treatment options with currently approved ARVs. | pregnancy, discontinuation of TMC125 development or when TMC125 has become commercially available in the patient's country.

SECONDARY OUTCOMES:
The secondary objective of this trial is to gather information on the safety and tolerability aspects of TMC125 in combination with other ARVs. Available efficacy data will also be collected. | pregnancy, discontinuation of TMC125 development or when TMC125 has become commercially available in the patient's country.

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Clinical Trial, Study Director — Tibotec Pharmaceutical Limited
Locations (259):
- United States (155):
  - Anniston, Alabama
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Tucson, Arizona
  - Anaheim, California
  - Arcata, California
  - Bakersfield, California
  - Beverly Hills, California
  - Fontana, California
  - Fountain Valley, California
  - Garden Grove, California
  - Harbor City, California
  - Hayward, California
  - Loma Linda, California
  - Long Beach, California
  - Los Angeles, California
  - Newport Beach, California
  - Oakland, California
  - Palm Springs, California
  - Panorama City, California
  - Sacramento, California
  - San Diego, California
  - San Francisco, California
  - San Mateo, California
  - San Rafael, California
  - Santa Ana, California
  - Santa Clara, California
  - Santa Clarita, California
  - Santa Rosa, California
  - Stanford, California
  - Tarzana, California
  - Ukiah, California
  - Woodland Hills, California
  - Denver, Colorado
  - Wheat Ridge, Colorado
  - Glastonbury, Connecticut
  - New Haven, Connecticut
  - Norwalk, Connecticut
  - Norwich, Connecticut
  - Washington D.C., District of Columbia
  - Daytona Beach, Florida
  - Fort Lauderdale, Florida
  - Fort Laudersale, Florida
  - Hollywood, Florida
  - LaBelle, Florida
  - Leesburg, Florida
  - Miami, Florida
  - North Miami Beach, Florida
  - North Palm Beach, Florida
  - Orlando, Florida
  - Pensacola, Florida
  - Plantation, Florida
  - Port Saint Lucie, Florida
  - Safety Harbor, Florida
  - Sarasota, Florida
  - Tampa, Florida
  - Tarpon Springs, Florida
  - Vero Beach, Florida
  - West Palm Beach, Florida
  - Winter Park, Florida
  - Atlanta, Georgia
  - Jesup, Georgia
  - Macon, Georgia
  - Riverdale, Georgia
  - Savannah, Georgia
  - Tucker, Georgia
  - Honolulu, Hawaii
  - Aurora, Illinois
  - Chicago, Illinois
  - Maywood, Illinois
  - Indianapolis, Indiana
  - Des Moines, Iowa
  - Iowa City, Iowa
  - Henderson, Kentucky
  - Paducah, Kentucky
  - New Orleans, Louisiana
  - Ellsworth, Maine
  - Portland, Maine
  - Baltimore, Maryland
  - Silver Spring, Maryland
  - Boston, Massachusetts
  - Springfield, Massachusetts
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Grand Rapids, Michigan
  - Grosse Pointe Woods, Michigan
  - Minneapolis, Minnesota
  - Rochester, Minnesota
  - Saint Louis Park, Minnesota
  - Kansas City, Missouri
  - St Louis, Missouri
  - Lincoln, Nebraska
  - Las Vegas, Nevada
  - Rochester, New Hampshire
  - Englewood, New Jersey
  - Hackensack, New Jersey
  - Long Branch, New Jersey
  - Neptune City, New Jersey
  - Newark, New Jersey
  - Perth Amboy, New Jersey
  - Somers Point, New Jersey
  - Voorhees Township, New Jersey
  - Westfield, New Jersey
  - Santa Fe, New Mexico
  - Briarcliff, New York
  - Brooklyn, New York
  - Buffalo, New York
  - East Meadow, New York
  - Elmira, New York
  - Flushing, New York
  - Kingston, New York
  - Manhasset, New York
  - New York, New York
  - Rochester, New York
  - Staten Island, New York
  - The Bronx, New York
  - Chapel Hill, North Carolina
  - Gastonia, North Carolina
  - Huntersville, North Carolina
  - Winston-Salem, North Carolina
  - Akron, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Dayton, Ohio
  - Portland, Oregon
  - Allentown, Pennsylvania
  - Johnstown, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Providence, Rhode Island
  - Columbia, South Carolina
  - Johnson City, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - El Paso, Texas
  - Fort Worth, Texas
  - Harlingen, Texas
  - Houston, Texas
  - Longview, Texas
  - San Antonio, Texas
  - Annandale, Virginia
  - Charlottesville, Virginia
  - Fairfax, Virginia
  - Hampton, Virginia
  - Norfolk, Virginia
  - Richmond, Virginia
  - Olympia, Washington
  - Seattle, Washington
  - Spokane, Washington
  - Yakima, Washington
  - Charleston, West Virginia
  - La Crosse, Wisconsin
  - Madison, Wisconsin
  - Milwaukee, Wisconsin
- Belgium (7):
  - Antwerp
  - Bruges
  - Brussels
  - Charleroi
  - Ghent
  - Leuven
  - Liège
- Canada (14):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Moncton, New Brunswick
  - Hamilton, Ontario
  - Kingston, Ontario
  - London, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Whitby, Ontario
  - Windsor, Ontario
  - Montreal, Quebec
  - Ste-Foy, Quebec
- Denmark (4):
  - Aarhus
  - Copenhagen
  - Hvidovre
  - Odense
- Germany (20):
  - Aachen
  - Berlin
  - Bochum
  - Bonn
  - Cologne
  - Düsseldorf
  - Erlangen
  - Essen
  - Frankfurt
  - Freiburg im Breisgau
  - Hamburg
  - Hanover
  - Mainz
  - Mannheim
  - Munich
  - München
  - Münster
  - Osnabrück
  - Stuttgart
  - Würzburg
- Greece (3):
  - Athens
  - Pátrai
  - Thessalonikis
- Luxembourg, Luxembourg
- Mexico (8):
  - Bosques Del Nogalar San Nicola
  - Chihuahua City
  - Col Tacuba
  - Guadalajara
  - Mexico City
  - Monterrey Nuevo León
  - Puebla City
  - Tijuana
- Netherlands (12):
  - Alkmaar
  - Amsterdam
  - Amsterdam-Zuidoost
  - Arnhem
  - Groningen
  - Leiden
  - Maastricht
  - Nijmegen
  - Rotterdam
  - The Hague
  - Tilburg
  - Utrecht
- San Juan, Puerto Rico
- Russia (3):
  - Moscow
  - Saint Petersburg
  - Volgograd
- South Korea (3):
  - Kyungki
  - Pusan
  - Seoul
- Spain (22):
  - Alicante
  - Barcelona
  - Bilbao
  - Cadiz
  - Cuenca
  - Elche
  - Granada
  - Granollers
  - Logroño
  - Madrid
  - Málaga
  - Murcia
  - Oviedo
  - Sabadell
  - San Cristóbal de La Laguna
  - Santa Cruz de Tenerife
  - Santiago de Compostela (La Cor
  - Seville
  - Terrassa
  - Valencia
  - Vigo
  - Vitoria-Gasteiz
- Sweden (3):
  - Gothenburg
  - Malmo
  - Stockholm
- Taiwan (2):
  - Kaohsiung City
  - Taipei
- Ankara, Turkey (Türkiye)

REFERENCES:
- See also: Early Access of TMC125 in Combination with Other Antiretrovirals in Treatment Experienced HIV-1 Infected Subjects with Limited Treatment Options — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=982&filename=CR002743_CSR.pdf